CLINICAL TRIAL: NCT05943717
Title: Lung Ultrasound Versus Cardiometry in Detection of Extravascular Lung Water in Pediatric Patients on Hemodialysis.
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sara Mabrouk Elghoul, Tanta, Stadium Street, Tanta University
Other Study IDs: 36264PR187/4/23
Record Dates: First submitted 2023-06-17; First posted 2023-07-13 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Fluid Volume Excess
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 50 children and adolescents with end stage renal disease on regular hemodialysis: 50 children and adolescents with end stage renal disease on regular hemodialysis for three times weekly
  Interventions: Device: lung ultrasound and electrical cardiometry

INTERVENTIONS:
Device: lung ultrasound and electrical cardiometry — : B-lines of lung ultrasound and the parameters of cardiometry will be measured at the mid-week HD session before starting the session by 30 min then every 30min during HD session for 180 min and then after the end of the session of HD by 30 min and then The specificity and sensitivity of both techniques will be compared to each other

SUMMARY:
Comparing the efficacy of both lung ultrasound and electrical cardiometry to detect the extravascular lung water and volume status in pediatric patients on regular hemodialysis and use them as non-invasive methods for early detection of hypervolemia or euvolemia even before appearance of clinical symptoms to decrease morbidity and mortality

DETAILED DESCRIPTION:
This cross sectional study will be conducted to compare between the efficacy of both lung ultrasound and electrical cardiometry to detect the extravascular lung water and volume status in pediatric patients on regular hemodialysis and use them as a non-invasive method for early detection of hypervolemia or euvolemia even before appearance of clinical symptoms of both conditions.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with end stage renal disease aged from 5 to 18 years on regular hemodialysis

Exclusion Criteria:

* Patients with coexisting lung fibrosis, atelectasis, and interstitial lung disease.
* Patients with heart failure.
* Patients with implantable cardiac pacemaker or defibrillator

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 50 children and adolescents with end stage renal disease on regular hemodialysis for three times weekly at TUH during the period of the study.
  Inclusion criteria: Pediatric patients with end stage renal disease aged from 5 to 18 years on regular hemodialysis.
  Exclusion criteria:
  * Patients with coexisting lung fibrosis, atelectasis, and interstitial lung disease.
  * Patients with heart failure.
  * Patients with implantable cardiac pacemaker or defibrillator.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
volume status in pediatric patients on regular hemodialysis | six months
  detection of the fluid status in pediatric patients on regular hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Sara Mabrouk Mohamed Elghoul, MD, Principal Investigator — Tanta University
Locations (1):
- Sara Mabrouk Mohamed Elghoul, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No